CLINICAL TRIAL: NCT02480725
Title: The Role of the Coagulation Pathway at the Synapse in Prion Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Prof. Zerr , Prion Referral Center , University of Gottingen, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. Oren Cohen, MD, Sheba Medical Center
Other Study IDs: 1702-14 SMC
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Creutzfeldt-Jakob Syndrome
Keywords: CJD; CSF; prion; thrombin
MeSH Terms: conditions — Creutzfeldt-Jakob Syndrome; Insomnia, Fatal Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CJD (Creutzfeldt-Jakob disease) patients: Prior to inclusion in the study a senior neurologist will interview the patient and will verify that he fully understands the objectives of the study and he is mentally qualified to sign the informed consent form (severely demented patients who will not be able to adequately consider the participation in the study will be excluded).
  Cognitive performance will be evaluated using the Mini-mental Status Examination and Frontal Assessment Battery scales.
  No clinical data other than the cognitive assessment and those needed for the clinical work up will be especially collected for this study.
  We plan to collect CSF samples for thrombin activity assay.
- non-CJD patients with a type of dementia: Prior to inclusion in the study a senior neurologist will interview the patient and will verify that he fully understands the objectives of the study and he is mentally qualified to sign the informed consent form (severely demented patients who will not be able to adequately consider the participation in the study will be excluded).
  Cognitive performance will be evaluated using the Mini-mental Status Examination and Frontal Assessment Battery scales.
  No clinical data other than the cognitive assessment and those needed for the clinical work up will be especially collected for this study.
  We plan to collect CSF samples for thrombin activity assay.
  Interventions: Procedure: collect CSF (Cerebrospinal fluid) sample
- CSF samples of non-CJD patient used as control: CSF samples : Thrombin activity will be assayed.

INTERVENTIONS:
Procedure: collect CSF (Cerebrospinal fluid) sample — collecting CSF samples for thrombin activity assay
  Groups: non-CJD patients with a type of dementia

SUMMARY:
The study hypothesis is that that the deleterious effect of prions on the brain may be mediated (at least partially) by activation of serine proteases involved in the coagulation system. If this is true, then measurement of the activity of the coagulation system may be a marker of disease onset (in at higher risk individuals such as E200K* carriers) and for disease progression or activity in affected individuals. In addition, modulation of the coagulation system activity may be a potential tool for therapeutic intervention.

*E200K- E200K mutation (Glu to Lys substitution) in the prion protein gene

DETAILED DESCRIPTION:
We plan to collect Cerebrospinal fluid (CSF) samples for thrombin activity assay in order to test whether there is a difference in thrombin activity in the CSF between CJD (Creutzfeldt-Jakob disease) and non-CJD patients. CSF samples will be obtained from two sources 1. Patients with familial or sporadic CJD and control patients with other neurodegenerative disorders (e.g. SDAT**, NPH) that will be evaluated in Sheba Medical Center 2. From our collaborating group of Prof. Zerr in the German Prion Referral Center at the University of Gottingen which has a collection of thousands of CSF samples from patients with familial and sporadic CJD as well as ideal controls with other degenerative brain disease.

The study has 2 sections:

1. Prospective part in which we plan to recruit 25 patients with CJD and 25 patients with other types of dementia from Sheba Medical Center (SMC). Prior to inclusion in the study a senior neurologist will interview the patient and will verify that he fully understands the objectives of the study and he is mentally qualified to sign the informed consent form (severely demented patients who will not be able to adequately consider the participation in the study will be excluded).

   Cognitive performance will be evaluated using the Mini-mental Status Examination and Frontal Assessment Battery scales.

   No clinical data other than the cognitive assessment and those needed for the clinical work up will be especially collected for this study.
2. Retrospective part in which CSF samples from CJD patients and patients with other type of dementia will be shipped to us from our collaborators in Germany ans will be assayed for Thrombin activity. We plan to recruit to this part of the study 100-200 CJD patient CSF samples and a same number of samples from age matched controls.

Thrombin activity (for samples from both parts of the study) will be assayed as follows: CSF sample will be placed in a black 96 well dish (10 per well). Thrombin activity will be measured by a fluorometric assay, quantifying the cleavage of the synthetic peptide substrate Boc-Asp(OBzl)-Pro-Arg-AMC*** (I-1560, Bachem, Switzerland, 13 molar final concentration). Measurements will be performed by the Infinite 2000 microplate reader (Tecan, infinite 200, Switzerland) with excitation and emission filters of 360±35 and 460±35 nm, respectively. CSF testing for thrombin activity will be conducted in Professor Chapman's laboratory in Sheba. This laboratory is actively engaged in research on the role of thrombin and PAR-1 in diseases of the nervous system and is fully equipped to perform the biochemical and protein levels experiments.

The assay has the potential for commercialization as a diagnostic test for CJD. In addition, there is the potential to develop therapeutic agents targeting excessive thrombin activation.

**SDAT=Senile Dementia of Alzheimer Type

***AMC= Amino Methyl Coumarin

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing lumbar puncture test as part of the investigation of cognitive decline.

Exclusion Criteria:

* Patients on anticoagulation or those who have contraindication for undergoing lumbar puncture.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CJD and non-CJD patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Thrombin activity assay | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Oren Cohen, Dr. (MD), Principal Investigator — Cheba Medical Center

REFERENCES:
- [Background] Prusiner SB. Molecular biology of prion diseases. Science. 1991 Jun 14;252(5012):1515-22. doi: 10.1126/science.1675487.
- [Background] Harris DA, Lele P, Snider WD. Localization of the mRNA for a chicken prion protein by in situ hybridization. Proc Natl Acad Sci U S A. 1993 May 1;90(9):4309-13. doi: 10.1073/pnas.90.9.4309. PMID 8483948
- [Background] Windl O, Dempster M, Estibeiro P, Lathe R. A candidate marsupial PrP gene reveals two domains conserved in mammalian PrP proteins. Gene. 1995 Jul 4;159(2):181-6. doi: 10.1016/0378-1119(95)00064-d. PMID 7622046
- [Background] Bueler H, Aguzzi A, Sailer A, Greiner RA, Autenried P, Aguet M, Weissmann C. Mice devoid of PrP are resistant to scrapie. Cell. 1993 Jul 2;73(7):1339-47. doi: 10.1016/0092-8674(93)90360-3. PMID 8100741
- [Background] Collinge J, Whittington MA, Sidle KC, Smith CJ, Palmer MS, Clarke AR, Jefferys JG. Prion protein is necessary for normal synaptic function. Nature. 1994 Jul 28;370(6487):295-7. doi: 10.1038/370295a0. PMID 8035877
- [Background] Tobler I, Gaus SE, Deboer T, Achermann P, Fischer M, Rulicke T, Moser M, Oesch B, McBride PA, Manson JC. Altered circadian activity rhythms and sleep in mice devoid of prion protein. Nature. 1996 Apr 18;380(6575):639-42. doi: 10.1038/380639a0. PMID 8602267
- [Background] Aucouturier P, Geissmann F, Damotte D, Saborio GP, Meeker HC, Kascsak R, Kascsak R, Carp RI, Wisniewski T. Infected splenic dendritic cells are sufficient for prion transmission to the CNS in mouse scrapie. J Clin Invest. 2001 Sep;108(5):703-8. doi: 10.1172/JCI13155. PMID 11544275
- [Background] Pan KM, Baldwin M, Nguyen J, Gasset M, Serban A, Groth D, Mehlhorn I, Huang Z, Fletterick RJ, Cohen FE, et al. Conversion of alpha-helices into beta-sheets features in the formation of the scrapie prion proteins. Proc Natl Acad Sci U S A. 1993 Dec 1;90(23):10962-6. doi: 10.1073/pnas.90.23.10962. PMID 7902575
- [Background] Ellis V, Daniels M, Misra R, Brown DR. Plasminogen activation is stimulated by prion protein and regulated in a copper-dependent manner. Biochemistry. 2002 Jun 4;41(22):6891-6. doi: 10.1021/bi025676g. PMID 12033920
- [Background] Epple G, Schleuning WD, Kettelgerdes G, Kottgen E, Gessner R, Praus M. Prion protein stimulates tissue-type plasminogen activator-mediated plasmin generation via a lysine-binding site on kringle 2. J Thromb Haemost. 2004 Jun;2(6):962-8. doi: 10.1111/j.1538-7836.2004.00675.x. PMID 15140132
- [Background] Fischer MB, Roeckl C, Parizek P, Schwarz HP, Aguzzi A. Binding of disease-associated prion protein to plasminogen. Nature. 2000 Nov 23;408(6811):479-83. doi: 10.1038/35044100. PMID 11100730
- [Background] Praus M, Kettelgerdes G, Baier M, Holzhutter HG, Jungblut PR, Maissen M, Epple G, Schleuning WD, Kottgen E, Aguzzi A, Gessner R. Stimulation of plasminogen activation by recombinant cellular prion protein is conserved in the NH2-terminal fragment PrP23-110. Thromb Haemost. 2003 May;89(5):812-9. PMID 12719777
- [Background] Deininger MH, Trautmann K, Magdolen V, Luther T, Schluesener HJ, Meyermann R. Cortical neurons of Creutzfeldt-Jakob disease patients express the urokinase-type plasminogen activator receptor. Neurosci Lett. 2002 May 10;324(1):80-2. doi: 10.1016/s0304-3940(02)00168-4. PMID 11983300
- [Background] Zerr I, Bodemer M, Kaboth U, Kretzschmar H, Oellerich M, Armstrong VW. Plasminogen activities and concentrations in patients with sporadic Creutzfeldt-Jakob disease. Neurosci Lett. 2004 Nov 23;371(2-3):163-6. doi: 10.1016/j.neulet.2004.08.063. PMID 15519749
- [Background] Almeida LM, Basu U, Khaniya B, Taniguchi M, Williams JL, Moore SS, Guan LL. Gene expression in the medulla following oral infection of cattle with bovine spongiform encephalopathy. J Toxicol Environ Health A. 2011;74(2-4):110-26. doi: 10.1080/15287394.2011.529061. PMID 21218340
- [Background] Chapman J. Coagulation in inflammatory diseases of the central nervous system. Semin Thromb Hemost. 2013 Nov;39(8):876-80. doi: 10.1055/s-0033-1357482. Epub 2013 Oct 9. PMID 24108468
- [Background] Maggio N, Shavit E, Chapman J, Segal M. Thrombin induces long-term potentiation of reactivity to afferent stimulation and facilitates epileptic seizures in rat hippocampal slices: toward understanding the functional consequences of cerebrovascular insults. J Neurosci. 2008 Jan 16;28(3):732-6. doi: 10.1523/JNEUROSCI.3665-07.2008. PMID 18199772
- [Background] Maggio N, Itsekson Z, Dominissini D, Blatt I, Amariglio N, Rechavi G, Tanne D, Chapman J. Thrombin regulation of synaptic plasticity: implications for physiology and pathology. Exp Neurol. 2013 Sep;247:595-604. doi: 10.1016/j.expneurol.2013.02.011. Epub 2013 Feb 27. PMID 23454608
- [Background] Maggio N, Cavaliere C, Papa M, Blatt I, Chapman J, Segal M. Thrombin regulation of synaptic transmission: implications for seizure onset. Neurobiol Dis. 2013 Feb;50:171-8. doi: 10.1016/j.nbd.2012.10.017. Epub 2012 Oct 25. PMID 23103417
- [Background] Shavit E, Beilin O, Korczyn AD, Sylantiev C, Aronovich R, Drory VE, Gurwitz D, Horresh I, Bar-Shavit R, Peles E, Chapman J. Thrombin receptor PAR-1 on myelin at the node of Ranvier: a new anatomy and physiology of conduction block. Brain. 2008 Apr;131(Pt 4):1113-22. doi: 10.1093/brain/awn005. Epub 2008 Feb 25. PMID 18299297
- [Background] Shavit E, Michaelson DM, Chapman J. Anatomical localization of protease-activated receptor-1 and protease-mediated neuroglial crosstalk on peri-synaptic astrocytic endfeet. J Neurochem. 2011 Nov;119(3):460-73. doi: 10.1111/j.1471-4159.2011.07436.x. Epub 2011 Sep 23. PMID 21854391
- [Background] Beilin O, Gurwitz D, Korczyn AD, Chapman J. Quantitative measurements of mouse brain thrombin-like and thrombin inhibition activities. Neuroreport. 2001 Aug 8;12(11):2347-51. doi: 10.1097/00001756-200108080-00013. PMID 11496108
- [Background] Beilin O, Karussis DM, Korczyn AD, Gurwitz D, Aronovich R, Hantai D, Grigoriadis N, Mizrachi-Kol R, Chapman J. Increased thrombin inhibition in experimental autoimmune encephalomyelitis. J Neurosci Res. 2005 Feb 1;79(3):351-9. doi: 10.1002/jnr.20270. PMID 15605378
- [Background] Beilin O, Karussis DM, Korczyn AD, Gurwitz D, Aronovich R, Mizrachi-Kol R, Chapman J. Increased KPI containing amyloid precursor protein in experimental autoimmune encephalomyelitis brains. Neuroreport. 2007 Apr 16;18(6):581-4. doi: 10.1097/WNR.0b013e328091c1e6. PMID 17413661
- [Background] Itzekson Z, Maggio N, Milman A, Shavit E, Pick CG, Chapman J. Reversal of trauma-induced amnesia in mice by a thrombin receptor antagonist. J Mol Neurosci. 2014 May;53(1):87-95. doi: 10.1007/s12031-013-0200-8. Epub 2013 Dec 19. PMID 24352712
- [Background] Bushi D, Chapman J, Katzav A, Shavit-Stein E, Molshatzki N, Maggio N, Tanne D. Quantitative detection of thrombin activity in an ischemic stroke model. J Mol Neurosci. 2013 Nov;51(3):844-50. doi: 10.1007/s12031-013-0072-y. Epub 2013 Jul 31. PMID 23900720
- [Background] Cohen OS, Prohovnik I, Korczyn AD, Ephraty L, Nitsan Z, Tsabari R, Appel S, Rosenmann H, Kahana E, Chapman J. The Creutzfeldt-Jakob disease (CJD) neurological status scale: a new tool for evaluation of disease severity and progression. Acta Neurol Scand. 2011 Dec;124(6):368-74. doi: 10.1111/j.1600-0404.2011.01489.x. Epub 2011 Feb 8. PMID 21303352
- [Background] Padilla D, Beringue V, Espinosa JC, Andreoletti O, Jaumain E, Reine F, Herzog L, Gutierrez-Adan A, Pintado B, Laude H, Torres JM. Sheep and goat BSE propagate more efficiently than cattle BSE in human PrP transgenic mice. PLoS Pathog. 2011 Mar;7(3):e1001319. doi: 10.1371/journal.ppat.1001319. Epub 2011 Mar 17. PMID 21445238
- [Background] Llorens F, Zafar S, Ansoleaga B, Shafiq M, Blanco R, Carmona M, Grau-Rivera O, Nos C, Gelpi E, Del Rio JA, Zerr I, Ferrer I. Subtype and regional regulation of prion biomarkers in sporadic Creutzfeldt-Jakob disease. Neuropathol Appl Neurobiol. 2015 Aug;41(5):631-45. doi: 10.1111/nan.12175. Epub 2015 Apr 30. PMID 25134744